CLINICAL TRIAL: NCT02353156
Title: Single Blind, Randomized Controlled, Multicenter Study to Evaluate the Efficacy and Convenience of Electronic Bidet With Very Low Force Flow Fountain System for Pain Control and Wound Healing After Operation for Anal Disease, Compared to Conventional Sitz Bath
Brief Title: Posthemorrhoidectomy Pain Management With Electronic Bidet or Sitz Bath
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Collaborators: Daehang Hospital (Other); Coway Co (Unknown)
Responsible Party: Principal Investigator, Kyu Joo Park, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-3144
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Hemorrhoid
Keywords: Hemorrhoidectomy; postoperative pain; Sitz bath; Electronic bidet
MeSH Terms: conditions — Hemorrhoids; Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electronic bidet (Experimental): Electronic bidet for 3min at early morning for 4 weeks after hemorrhoidectomy
  Interventions: Other: Electronic bidet
- Sitz bath (Active Comparator): Wamr sitz bath for 3min at early morning for 4 weeks after hemorrhoidectomy
  Interventions: Other: Sitz bath

INTERVENTIONS:
Other: Electronic bidet — electronic bidet after hemorrhoidectomy for relieving pain and inducing wound healing
  Arms: Electronic bidet
Other: Sitz bath — sitz bath after hemorrhoidectomy for relieving pain and inducing wound healing
  Arms: Sitz bath

SUMMARY:
The investigator will perform a randomized clinical trials to compare the effect of pain management and wound healing after hemorrhoidectomy between warm sitz bath and electronic bidet.

DETAILED DESCRIPTION:
After hemorrhoidectomy, the patients should take warm sitz bath for relieving pain and inducing wound healing. Electronic bidet is a device for cleansing the anus after defecation, and some patients are using the bidet for sitz bath. Thus, the investigator perform this study for comparing the effect of pain and wound management after hemorrhoidectomy between sitz bath and electronic bidet

ELIGIBILITY:
Inclusion Criteria:

* the patients who undergo hemorrhoidectomy

Exclusion Criteria:

* previous history of anal surgery
* Crohn's anal disease
* perianal complex abscess or fistula
* uncontrollable medical disease
* Tb
* HIV
* malignancy
* immunocompromised
* pregnancy
* breast feeding
* NSAID allergy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
pain score | 1 week
  visual analog scale after hemorrhoidectomy at 1 week

SECONDARY OUTCOMES:
wound healing | 4 week
  wound healing rate at 4 week
convenience | 4 week
  questionnaire survey for convenience of wound management after hemorrhoidectomy
urinary difficulty | 4 week
  IPSS, urinary difficulty questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Joo Park, MD, PhD, Principal Investigator — Seoul National University College of Medicine

REFERENCES:
- [Background] Ryoo S, Song YS, Seo MS, Oh HK, Choe EK, Park KJ. Effect of electronic toilet system (bidet) on anorectal pressure in normal healthy volunteers: influence of different types of water stream and temperature. J Korean Med Sci. 2011 Jan;26(1):71-7. doi: 10.3346/jkms.2011.26.1.71. Epub 2010 Dec 22. PMID 21218033
- [Derived] Kwon YH, Ryoo SB, Oh HK, Lee JB, Jung HJ, Song KH, Heo SC, Shin R, Lee J, Park KJ. Comparison of warm sitz bath and electronic bidet with a lower-force water flow for postoperative management after hemorrhoidectomy (BIDLOW). BMC Surg. 2025 Jan 6;25(1):5. doi: 10.1186/s12893-024-02737-0. PMID 39757160